CLINICAL TRIAL: NCT04897503
Title: Randomized Study of Safety and Effectiveness of Corneal Collagen Crosslinking Using Riboflavin/Dextran or Riboflavin/Methylcellulose
Brief Title: Corneal Collagen Crosslinking for Keratoconus and Ectasia Using Riboflavin/Dextran or Riboflavin/Methylcellulose
Acronym: CXL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEI - ISO-CXL-001
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: keratoconus; corneal ectasia; collagen crosslinking; riboflavin; cornea; ultraviolet; crosslinking; corneal crosslinking
MeSH Terms: conditions — Keratoconus; Corneal Diseases | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CXL using Riboflavin/Dextran solution (Active Comparator): Corneal collagen crosslinking using 0.1% riboflavin mixed with 20% dextran
  Interventions: Drug: Riboflavin
- CXL usinng Riboflavin/Methylcellulose solution (Active Comparator): Corneal collagen crosslinking using 0.1% riboflavin mixed with 1.0% hydroxypropylmethylcellulose ( HPMC)
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Corneal epithelium removed followed by riboflavin drop administration (riboflavin/dextran -vs- riboflavin/methylcellulose) every 2 minutes for 30 minutes followed by UV light exposure with additional riboflavin administration every 2 minutes for 30 minutes. Subjects will be randomized to receive either the riboflavin/dextran solution or the riboflavin/HPMC solution.

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of isotonic riboflavin for corneal collagen crosslinking for keratoconus and corneal ectasia. will determine the safety and efficacy of corneal collagen crosslinking (CXL) performed with two different riboflavin formulations for reducing corneal curvature.

DETAILED DESCRIPTION:
This study will determine the safety and efficacy of corneal collagen crosslinking (CXL) performed with two different riboflavin formulations for reducing corneal curvature. Subjects will be randomized to one of 2 groups. One group will be treated with a methylcellulose riboflavin solution and the other group will be treated with a dextran riboflavin solution. Both groups will be exposed to 3mW/cm2 of continuous UVA light for a total of 30 minutes; each group will continue to be administered the designated riboflavin drops during UV exposure.

The primary efficacy parameter that will be evaluated over time is maximum keratometry (Kmax) in the randomized eyes for each treatment group.

The secondary efficacy parameter will be to determine if the two treatment groups equivalent in their Kmax change at 12 months after treatment compared with baseline.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Having a diagnosis of keratoconus or corneal ectasia after corneal refractive surgery
* Presence of central or inferior steepening on the Pentacam map
* Axial topography consistent with keratoconus or post-surgical corneal ectasia
* Contact lens wearers only: removal of contact lens for the required period of 1 week prior to the screening refraction
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme
* Corneal pachymetry less than or equal to 300 microns at the thinnest point measured by Pentacam in the eye(s) to be treated
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications, for example: History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.) Clinically significant corneal scarring in the CXL treatment zone
* A history of chemical injury or delayed epithelial healing in the eye(s) to be treated
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum keratometry | 12 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 12 months for all eyes randomized in group 1 and group 2.

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Change in uncorrected visual acuity (UCVA) and best spectacle corrected visual acuity (BCVA) compared to the baseline examination will be evaluated at 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hersh, MD, Study Director — Cornea and Laser Eye Institute Hersh Vision Group; Steven A Greenstein, MD, Principal Investigator — Cornea and Laser Eye Institute, Hersh Vision Group
Locations (1):
- Cornea and Laser Eye Institue - Hersh Vision Group, Teaneck, New Jersey, United States